CLINICAL TRIAL: NCT05360641
Title: Risk Factors for Recurrence of Thrombosis or Thrombotic Extension, in the Event of Acute Non-cirrhotic Portal Vein Thrombosis Secondary to a Local Cause.
Acronym: LOCAPORT
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAPORT
Record Dates: First submitted 2022-04-12; First posted 2022-05-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2022-04

CONDITIONS: Portal Vein Thrombosis; Local Cause
Keywords: liver vascular disease; portal vein thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In case of acute portal vein thrombosis (PVT) prothrombotic factors are identified in about 60% of cases, while a local condition is present in 30% of cases. Prothrombotic factors may indicate a long term anticoagulant therapy whereas the risk of recurrence seems low when a local condition is isolated (cholecystitis, angiocholitis, liver abces, diverticulitis, appendicitis, acute/chronic pancreatitis, chronic bowel inflammatory disease, acute hepatitis due to cytomegalovirus, bacteroïdes pylephlebitis, abdominal neoplasia such as adenocarcinoma of the colon, abdominal traumatism or surgery such as cholecystectomy, bariatric surgery or splenectomy). To date the impact of prothrombotic factors associated with local conditions responsible for acute PVT has not been well studied except for acute or chronic pancreatitis. No significant association has been pointed out in this pathology. The aim is to determine what are the risk factors of thrombotic recurrence or extension associated with local conditions responsible for acute non cirrhotic PVT, and to evaluate the rate of secondary long term anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* acute portal thrombosis segmental or truncal, diagnosed in the context of a local inflammatory, infectious, trauma or abdominal surgery cause, dating from less than 3 months.
* patients already included in european cohort ENVIE-VALDIG

Exclusion Criteria:

* liver cirrhosis
* liver, biliary or pancreatic neoplasia
* thrombosis limited to mesenteric vein, splenic vein or splenomesaraic confluence
* cavernoma or Budd-Chiari syndrom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years of age or older with acute portal thrombosis segmental or truncal diagnosed in the context of a local cause inflammatory, infectious, trauma or abdominal surgery dating from less than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of thrombosis at 5 years | 5 years
  Risk factor for recurrence of thrombosis at 5 years (regardless of territory), or splanchnic thrombotic extension, in case of acute non-cirrhotic PVT secondary to a local cause of infection, inflammation, trauma or abdominal surgery.

SECONDARY OUTCOMES:
Prevalence of thrombotic factors | 5 years
  Prevalence of thrombotic factors with its 95% confidence interval.
Prothrombotic factors | 5 years
  Interest of a systematic search for prothrombotic factors in terms of prevention of recurrence of thrombosis, mortality (morbidity, mortality)
Long-term anticoagulation | 5 years
  Percentage of indications for long-term anticoagulation at the end of the exhaustive search for prothrombotic factors: this percentage will be estimated with its IC 95

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Caen, Caen, Calvados, France